CLINICAL TRIAL: NCT06952465
Title: A Cohort Study Comparing the Risk of Serious Infections and Malignancies With Deucravacitinib or Biologics in Japanese Patients With Plaque Psoriasis, Generalized Pustular Psoriasis, and Erythrodermic Psoriasis Using Administrative Health Claims Database
Brief Title: A Study Comparing the Risk of Serious Infections and Malignancies With Deucravacitinib or Biologics in Japanese Patients With Psoriasis
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-227
Record Dates: First submitted 2025-04-29; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis
Keywords: Psoriasis (PsO)
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Cohort 1: Participants receiving deucravacitinib treatment
  Interventions: Drug: Deucravacitinib
- Cohort 2: Participants receiving biologics treatment for psoriasis
  Interventions: Biological: Any biologic treatment for psoriasis

INTERVENTIONS:
Drug: Deucravacitinib — As per product label
  Groups: Cohort 1
Biological: Any biologic treatment for psoriasis — According to the product label
  Groups: Cohort 2

SUMMARY:
The purpose of this study is to further evaluate the safety of deucravacitinib treatment in Japanese patients with psoriasis in the real-world setting

ELIGIBILITY:
Inclusion Criteria:

* Participants with prescriptions in deucravacitinib or any biologics as comparator group during the indexing period.
* Participants with at least one confirmed diagnosis of disease code for psoriasis within 12 months prior to the index date.
* Aged 18 years or older at the index date

Exclusion Criteria:

* Participants with prescription in deucravacitinib or any biologics as comparator group prior to the index date.
* Participants with fewer than 12 months of available claim records prior to the index date.
* Participants with no claims record within 1-year after the index date (no visit after the index date).
* Specific for serious infection: Participants who had at least one disease code of hospitalized infection in the 60 days period before the index date.
* Specific for malignancy: Participants who had at least one disease code of malignancy prior to the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients identified from the Japanese healthcare claims database with psoriasis who have initiated either deucravacitinib or any biologic treatment for psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2031-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Participant baseline demographics | Baseline
Participant medical history | Baseline
Incidence of serious infections | Up to 9-years
Incidence of malignancies | Up to 9-years

SECONDARY OUTCOMES:
Incidence of serious infections excluding COVID-19 | Up to 9-years
Incidence of serious infection of COVID-19 | Up to 9-years
Incidence of opportunistic infections excluding tuberculosis and herpes zoster | Up to 9-years
Incidence of tuberculosis | Up to 9-years
Incidence of herpes zoster | Up to 9-years
Incidence of malignancies excluding non-melanoma skin cancer | Up to 9-years
Incidence of non-melanoma skin cancer | Up to 9-years
Incidence of solid tumors | Up to 9-years
Incidence of hematologic malignancies | Up to 9-years
Incidence of lymphoma | Up to 9-years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Local Institution, Tokyo
  - Medical Data Vision, Inc, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm